CLINICAL TRIAL: NCT00921544
Title: Sucrose and Non Nutritive Suck as Analgesia for Babies Undergoing Retinopathy of Prematurity Screening; a Randomised Placebo Controlled Trial
Brief Title: Sucrose Analgesia for the Reduction of Pain During Retinopathy of Prematurity Screening
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coombe Women and Infants University Hospital (Other)
Responsible Party: Eugene Dempsey, Coombe Women and Infants University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Coombesucrose
Record Dates: First submitted 2009-06-10; First posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Retinopathy of Prematurity
Keywords: ROP; sucrose; pain
MeSH Terms: conditions — Retinopathy of Prematurity; Pain | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Sucrose (Active Comparator): Oral sucrose administered 2 mins prior to eye exam
  Interventions: Other: Sucrose
- Sterile water (Placebo Comparator): 0.2 mls of sterile water
  Interventions: Other: Sterile water

INTERVENTIONS:
Other: Sucrose — 0.2 ml sucrose 24% given by mouth using a syringe and pacifier
  Other Names: Sweeties
  Arms: Oral Sucrose
Other: Sterile water — Sterile water administered 2 mins prior to eye exam
  Arms: Sterile water

SUMMARY:
Retinopathy of Prematurity (ROP) screening is one of many potentially painful diagnostic and therapeutic procedures performed routinely on preterm infants in the Neonatal Intensive Care Unit. Therefore strategies for stress reduction and pain management are essential to promote growth and development and minimize long-term sequelae. Procedural analgesia should include concepts of developmental care, non nutritive suck (NNS), pharmacological and non-pharmacological agents. Sucrose is thought to stimulate the body's activation of lingual sweet taste receptors and release of endogenous opioids, when combined with NNS, non-opioid mechanisms are also activated. The administration of sucrose or the combination of sucrose and non-nutritive sucking is one of the most frequently studied non-pharmacological interventions for relief of pain in neonates and oral sucrose has been shown to be an effective and safe therapy for common neonatal procedures such as heal lance, blood-letting and venepuncture. There is conflicting evidence on the benefit of sucrose in ROP screening. Therefore the purpose of this study is to determine the efficacy of sucrose combined with NNS as a potential regime for reduction of pain associated with retinopathy of prematurity screening.

ELIGIBILITY:
Inclusion Criteria:

* < 1500 grams
* < 32 weeks

Exclusion Criteria:

* Requiring mechanical ventilation excluding Continuous Positive Pressure Ventilation (CPAP), sedation
* Infants where consent to participate was not obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pain profile score as assessed by NPASS | Scores assessed 3 months following completion of study

SECONDARY OUTCOMES:
Number of adverse events | Assessed 3 months following completion

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Dempsey, MD, FRCPI, Study Director — Coombe Women and Infants University Hospital
Locations (1):
- Coombe Women and Infants University Maternity Hospital, Dublin, Dublin, Ireland